CLINICAL TRIAL: NCT00481897
Title: Worksite Nutrition Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCCR-07065-01
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Overweight; Type 2 Diabetes
Keywords: overweight; obesity; type 2 diabetes; diabetes; worksite cost; nutrition
MeSH Terms: conditions — Overweight; Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus | interventions — Diet, Fat-Restricted; Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: low-fat, vegan diet — Diet that excludes animal products (i.e. meat, dairy, eggs) and keeps oils to a minimum.

SUMMARY:
The Worksite Nutrition Study is 22-week translational study aimed at determining how well a worksite-based nutrition program, as compared to a control group, is able to 1) produce clinically significant weight-loss, 2) improve cardiovascular factors, 3) decrease work absenteeism, 4) improve overall quality of life, 5) improve diabetes control in participants with diabetes, and 6) promote dietary adherence and acceptability. The nutrition program for the intervention group consists of once-weekly group meetings where participants will receive group support and nutrition education on a low-fat, vegan diet.

DETAILED DESCRIPTION:
Approximately 65 percent of Americans are overweight or obese. They are at increased risk for diabetes, hypertension, dyslipidemia, cardiovascular disease, arthritis, respiratory disorders, pregnancy complications, and premature death. Research has demonstrated that weight status is associated with certain types of malignancies, including endometrial, colon, gall bladder, prostate, kidney, and postmenopausal breast cancer. The total direct and indirect costs attributed to overweight and obesity amounted to 117 billion U.S. dollars in 2000.

The 22-week Worksite Nutrition Study will (1) test whether a worksite intervention, which prescribes a low-fat vegan diet, is effective in promoting clinically significant weight loss, (2) evaluate whether the intervention reduces cardiovascular risk, particularly blood pressure and lipid concentrations, (3) assess whether the intervention improves glycemic control in individuals with type 2 diabetes, and (4) examine how the intervention affects work impairment and absenteeism.

Participants (Group 1, n=60) at a specified worksite will be assigned to the diet intervention program, which prescribes a low-fat, vegan diet. A control group (Group 2, n=60) will be designated at a separate worksite. The participants in the control group will not receive an active intervention during the designated study period. Participants in the active intervention will attend weekly group meetings for nutrition education on the intervention diet.

Diets will be assessed, in order to monitor adherence and for the purposes of comparison, in the intervention and control groups at baseline and at weeks 11 and 22 using a 3-day dietary record. Dependent measures, including body weight, blood pressure, lipid concentrations, quality-of-life measures, and A1c (for those with diabetes) will be assessed in the intervention and control groups at weeks 0, 11, and 22.

ELIGIBILITY:
Inclusion Criteria:

* employee at the intervention worksite or the control worksite;
* BMI > 25 or a diagnosis of type 2 diabetes mellitus, as defined by a fasting plasma glucose concentration > 126 mg/dl on two occasions or a prior physician's diagnosis of type 2 diabetes with the use of hypoglycemic medications for at least six months;
* male or female;
* age at least 18 years;
* ability and willingness to participate in all components of the study; and
* a willingness to be assigned to a low-fat, vegan diet or control group.

Exclusion Criteria:

* a history of alcohol abuse or dependency followed by any current use;
* current or unresolved past drug abuse;
* pregnancy;
* history of severe mental illness;
* unstable medical status;
* already following a low-fat, vegetarian diet;
* an inordinate fear of blood draw; and
* A1c <7 or >10.5% (for volunteers with diabetes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Assignment to a diet intervention program promotes clinically significant weight loss, compared to a control group. | 22 weeks
Assignment to the diet intervention program improves indices of cardiovascular risk, including plasma lipid concentrations and blood pressure, compared to a control group. | 22 weeks
Assignment to the diet intervention program improves glycemia in a sub-group of participants with type 2 diabetes, as indicated by mean A1c, relative to matched participants with type 2 diabetes in the control group. | 22 weeks
Assignment to the diet intervention, decreases the prevalence of work absenteeism, as measured by the proportion of days that a participant is absent from work, compared with assignment to a control group. | 22 weeks

SECONDARY OUTCOMES:
Assignment to the diet intervention improves quality of life measures, including general mental and physical health, relative to assignment to a control group. | 22 weeks
Assignment to the diet intervention program promotes adherence and acceptability. | 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hope Ferdowsian, M.D., M.P.H., Principal Investigator — Washington Center for Clinical Research; Neal Barnard, M.D., Principal Investigator — Washington Center for Clinical Research
Locations (1):
- Washington Center for Clinical Research, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Levin SM, Ferdowsian HR, Hoover VJ, Green AA, Barnard ND. A worksite programme significantly alters nutrient intakes. Public Health Nutr. 2010 Oct;13(10):1629-35. doi: 10.1017/S136898000999303X. Epub 2010 Jan 15. PMID 20074388
- [Result] Katcher HI, Ferdowsian HR, Hoover VJ, Cohen JL, Barnard ND. A worksite vegan nutrition program is well-accepted and improves health-related quality of life and work productivity. Ann Nutr Metab. 2010;56(4):245-52. doi: 10.1159/000288281. Epub 2010 Apr 14. PMID 20389060
- [Result] Ferdowsian HR, Barnard ND, Hoover VJ, Katcher HI, Levin SM, Green AA, Cohen JL. A multicomponent intervention reduces body weight and cardiovascular risk at a GEICO corporate site. Am J Health Promot. 2010 Jul-Aug;24(6):384-7. doi: 10.4278/ajhp.081027-QUAN-255. PMID 20594095